CLINICAL TRIAL: NCT00010829
Title: Macrobiotic Diet and Flax Seed: Effects on Estrogens, Phytoestrogens, & Fibrinolytic Factors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: P50AT000090-01P1 (NIH); P50AT000090-01 (NIH); NCT00009425 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Cardiovascular Diseases; Osteoporosis; Breast Cancer; Endometrial Cancer
Keywords: Cardiovascular Diseases; Osteoporosis; Breast Cancer; Endometrial Cancer
MeSH Terms: conditions — Cardiovascular Diseases; Osteoporosis; Breast Neoplasms; Endometrial Neoplasms | interventions — Linseed Oil

INTERVENTIONS:
Behavioral: American Heart Association Step 1 diet
Behavioral: American Heart Association Step 2 diet + 10 g/day flax seed
Behavioral: Macrobiotic dietary intervention

SUMMARY:
This study will assess whether alternative, high phytoestrogen dietary interventions result in favorable effects on biological parameters that have been associated with hormone-dependent cancers, cardiovascular disease, and osteoporosis.

DETAILED DESCRIPTION:
Broad health effects of endogenous and exogenous estrogens on diseases of aging, including hormone-dependent cancers, cardiovascular disease, and osteoporosis, are generally recognized. For example, estrogen replacement therapy (ERT) may increase the risk of subsequent breast and endometrial cancer, but also decreases the risk of coronary disease and fractures. Because of the increased cancer risk, many women seek out alternatives to ERT. Phytoestrogens, plant compounds that have estrogenic effects, have been a focus of interest as an alternative to ERT. The isoflavones and lignans are two major classes of phytoestrogens that occur in the food supply. Among the former, soy foods have attracted much interest, while among the latter, whole grains and seeds are sources in a typical diet. More specifically, women consuming a macrobiotic diet have been observed to have extremely high levels of phytoestrogen metabolites in their urine, perhaps 10 to 20 times that seen in women consuming an omnivorous diet. Proponents of a macrobiotic diet have proposed that it is beneficial in the context of cancer therapy, as well as for the prevention and treatment of cardiovascular disease.

This study will investigate, in a randomized, three-arm study, the effects of two interventions that are high in phytoestrogens on various parameters related to estrogen metabolism and fibrinolysis. Approximately 120 women will be randomized to receive an American Heart Association (AHA) Step 1 diet, an AHA Step 2 diet + 10 g/day flax seed, or a macrobiotic dietary intervention. Blood and urine samples will be drawn at baseline, and at three, six, nine, and twelve months, to examine both short and long-term effects of these interventions. Outcomes include blood and urine levels of total estrogens and estradiol, and related metabolites; antigens to plasminogen activator inhibitor-1 (PAI-1) and tissue plasminogen activator (t-PA), fibrin D-dimer, and von Willebrand Factor; and endothelial function as measured by high-resolution ultrasound. Blood levels of antioxidant vitamins and retinoids will also be examined.

This study should provide information on whether these alternative, high phytoestrogen dietary interventions result in favorable effects on these biological parameters that are related to risk of major diseases of aging.

ELIGIBILITY:
Inclusion Criteria:

THIS TRIAL IS RECRUITING IN THE NEW YORK METRO AREA ONLY

* Postmenopausal
* Weight within 90% to 120% of ideal body weight

Ages: 50 Years to 72 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2001-01; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Lawrence Kushi, Principal Investigator — Columbia University, Teachers College
Locations (1):
- Columbia University, New York, New York, United States